CLINICAL TRIAL: NCT02408224
Title: A Non-interventional Prospective Observational Study to Understand the Usage Pattern of Ticagrelor in Indian Patients With Acute Coronary Syndrome.
Brief Title: An Observational Prospective Study to Understand the Usage Pattern of Ticagrelor With ACS (Acute Coronary Syndrome)
Acronym: TREASURE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130R00029; NIS-CIN-BRI-2014/1 (Other: AstraZeneca)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one arm: patients on Ticagrelor

SUMMARY:
The TREASURE observational study is designed to address the need to understand the usage pattern of Ticagrelor in real life scenario in large number of ACS (Acute Coronary Syndrome) patients in India. The aim of this national study is to understand the usage pattern (including the duration of treatment) of Ticagrelor in various ACS patient population undergoing PCI (Percutaneous Coronary Intervention), CABG (Coronary Artery Bypass Graft) or medical management in a real-life setting in India.

DETAILED DESCRIPTION:
This study is a multi-centre, observational, prospective study to be conducted at 60 hospitals across IndiaThe study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) and written Informed consent of the patient.

Patients who had been hospitalized for ACS and are on ticagrelor on discharge or on Ticagrelor therapy for ≤ 1month will be enrolled in the study and followed up for a period of 12 months. During the follow-up period of up to 12 months (according to the label), assessment visits will follow the routine clinical practice. No visits or measurements will be made mandatory by the protocol

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been provided.
2. Aged 18 years or older.
3. Male/female with ACS on Ticagrelor on discharge or ≤ 1month.
4. Patient underwent PCI, CABG or MM (Medical Management) for ACS.
5. Diagnosis of STEMI, NSTEMI or UA

Exclusion Criteria:

1. Patients with medical history of intracranial hemorrhage
2. All those patients who are not fit to receive Ticagrelor as per the latest prescribing information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male/female with Acute Coronary Syndrome on Ticagrelor on discharge or ≤ 1month
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2017-06-24 (Actual); Study Completion 2017-06-24 (Actual)

PRIMARY OUTCOMES:
Usage pattern of Ticagrelore in real life setting | 48 Weeks
  Assessing the proportion of enrolled patients with different types of ACS namely, STEMI (ST segment Elevation Myocardial Infarction), NSTEMI (Non-ST segment Elevation Myocardial Infarction) and UA (Unstable Angina)
Usage pattern of Ticagrelore | 48 Weeks
  Assessing the proportion of patients with different types of ACS management namely, PCI, CABG and Medical Management

SECONDARY OUTCOMES:
Frequency of various risk factors | 48 Weeks
  GRACE (Global Registry of Acute Coronary Events) score

CONTACTS AND LOCATIONS:
Overall Officials: JP S Sawhney, MBBS, MD, DM, Study Chair — Sir Ganga Ram Hospital, Delhi; Bhavesh P Kotak, MBBS MD, Study Director — AstraZeneca Pharma India Ltd
Locations (31):
- India (31):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Vijayawada, Andhra Pradesh
  - Research Site, Patna, Bihar
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Surat, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Gurgaon, Haryana
  - Research Site, Srinagar, Jammu and Kashmir
  - Research Site, Bangalore, Karnataka
  - Research Site, Bengaluru, Karnataka
  - Research Site, Mysore, Karnataka
  - Research Site, Kolenchery, Kerala
  - Research Site, Thrissur, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Delhi, New Delhi
  - Research Site, Bhubaneswar, Odisha
  - Research Site, Ludhiana, Punjab
  - Research Site, Mohali, Punjab
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Hyderabad, Telangana
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Noida, Uttar Pradesh
  - Research Site, Durgapur, West Bengal
  - Research Site, Kolkata, West Bengal

REFERENCES:
- [Derived] Sawhney JPS, Dalal J, Mullasari A, Bansal S, Kahali D. Therapeutic experience of ticagrelor in Indian patients with acute coronary syndrome: A non-interventional, prospective, and observational study. Indian Heart J. 2019 Jul-Aug;71(4):344-349. doi: 10.1016/j.ihj.2019.08.001. Epub 2019 Aug 30. PMID 31779864
- See also: Revised CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3820&filename=TREASURE%20CSR_Synopsis%20revised%20FINAL.pdf